CLINICAL TRIAL: NCT07399041
Title: A Prospective Single-Center Study Evaluating the Effects of Adenoidectomy and Adenotonsillectomy on Voice and Speech Functions in Children
Brief Title: Evaluation of the Effects of Adenoidectomy and Adenotonsillectomy on Voice in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ENT-PROS-AD-AT-2026
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Adenoid Hypertrophy; Tonsillar Hypertrophy; Voice Disorders in Children
Keywords: Adenoidectomy; Adenotonsillectomy; Pediatric Voice; Nasalance; praat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children Undergoing Adenoidectomy or Adenotonsillectomy: Children aged 4-13 years scheduled for routine adenoidectomy or adenotonsillectomy. Participants are followed prospectively to evaluate changes in voice and speech parameters before surgery and at postoperative 1st and 3rd months.

SUMMARY:
This prospective study aims to evaluate the effects of adenoidectomy and adenotonsillectomy on voice and speech functions in children. Changes in voice quality and resonance may occur after the removal of adenoid and tonsillar tissues, particularly in pediatric patients with enlarged adenoids or tonsils.

Objective voice assessments, including acoustic, aerodynamic, and nasalance measurements, as well as subjective voice-related quality of life questionnaires, will be performed before surgery and at the first and third months after surgery. The results of this study are expected to help clinicians better inform families about possible voice changes following adenoidectomy and adenotonsillectomy procedures.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study designed to evaluate the effects of adenoidectomy and adenotonsillectomy on voice and speech functions in pediatric patients.

A minimum of 36 children aged between 4 and 13 years who are scheduled for primary adenoidectomy or adenotonsillectomy will be included in the study. Written informed consent will be obtained from the parents or legal guardians of all participants prior to enrollment. All patients will undergo routine otolaryngological examination.

Voice recordings will be obtained in a sound-isolated room one day before surgery and at the first and third postoperative months. Recordings will be performed using an AKG P5-S dynamic microphone (AKG®, Vienna, Austria) and a Behringer UMC22 audio interface (Behringer®, Willich, Germany). The microphone will be positioned at approximately a 90-degree angle and 10 cm from the mouth while the patient is seated.

Participants will be instructed to sustain the vowel /a/ at a comfortable pitch and loudness following deep inspiration, repeated three times. The longest sustained phonation will be recorded as the maximum phonation time and used as an aerodynamic parameter.

Acoustic analysis will be performed using Praat software (Version 6.1.39; Paul Boersma and David Weenink, University of Amsterdam). Sustained vowel samples of 3-5 seconds will be analyzed to obtain fundamental frequency (F0), jitter, shimmer, and harmonics-to-noise ratio (HNR) values.

Nasalance measurements will be conducted using a Plex device and a dynamic microphone to evaluate nasal resonance and determine whether resonance values fall within normal limits.

All voice recordings will be captured using Audacity software and analyzed using Praat. Subjective voice assessment will be performed using the Pediatric Voice Handicap Index and the Pediatric Voice-Related Quality of Life questionnaires, both of which have been validated in Turkish. These questionnaires will be administered preoperatively and at the first and third postoperative months.

The study aims to provide objective and subjective data regarding voice changes following adenoidectomy and adenotonsillectomy and to support preoperative counseling of families regarding potential postoperative voice outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4-13 years
* Scheduled for primary adenoidectomy or adenotonsillectomy

Exclusion Criteria:

* Does not meet inclusion criteria
* Refuses to participate in the study
* Diagnosis of vocal cord disorders
* History of vocal cord surgery
* History of cleft palate or cleft lip
* Hearing loss requiring a hearing aid
* Chronic diseases that may impair wound healing, including: hypertension, diabetes mellitus, immunodeficiency, autoimmune diseases, rheumatologic diseases, connective tissue disorders, renal failure, liver failure, chronic heart disease
* Known bleeding diathesis
* Use of anticoagulant or antiplatelet drugs
* Upper respiratory tract infection within the last 2 weeks
* Patients undergoing revision adenoidectomy

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study includes children aged 4-13 years who are scheduled for primary adenoidectomy or adenotonsillectomy. The aim is to evaluate the effects of these surgical procedures on voice and speech function, using both objective acoustic measurements and validated pediatric voice-related quality of life questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Fundamental Frequency (F0) | Preoperative, 1 month postoperative, and 3 months postoperative
  Fundamental frequency (F0), expressed in Hertz (Hz), will be measured using objective acoustic voice analysis with Praat software. Measurements will be obtained from sustained vowel /a/ recordings and compared between preoperative and postoperative evaluations.
Change in Jitter Percentage | Preoperative, 1 month postoperative, and 3 months postoperative
  Jitter, expressed as a percentage (%), will be measured from sustained vowel /a/ recordings using Praat software. Preoperative jitter values will be compared with postoperative measurements at the 1st and 3rd months to assess changes in frequency stability after surgery.
Change in Shimmer Percentage | Preoperative, 1 month postoperative, and 3 months postoperative
  Shimmer, expressed as a percentage (%), will be measured from sustained vowel /a/ recordings using Praat software. Measurements obtained preoperatively will be compared with postoperative values at the 1st and 3rd months to evaluate changes in amplitude stability following surgery.
Change in Harmonics-to-Noise Ratio (HNR) | Preoperative, 1 month postoperative, and 3 months postoperative
  Harmonics-to-noise ratio (HNR), measured in decibels (dB), will be obtained from sustained vowel /a/ recordings using Praat software. Preoperative and postoperative (1st and 3rd months) values will be compared to assess changes in voice signal quality after surgery.

SECONDARY OUTCOMES:
Change in Nasalance Scores After Surgery | Preoperative, 1 month postoperative, and 3 months postoperative
  Nasalance will be measured using a nasalance measurement system with a plex device and dynamic microphone. Nasalance scores are expressed as percentages ranging from 0% to 100%, with higher scores indicating increased nasal resonance. Preoperative and postoperative measurements will be compared.
Change in Pediatric Voice Handicap Index Scores | Preoperative, 1 month postoperative, and 3 months postoperative
  Subjective voice outcomes will be assessed using the Pediatric Voice Handicap Index (PVHI). The total score ranges from 0 to 92, with higher scores indicating greater perceived voice-related handicap. The validated Turkish version of the questionnaire will be administered preoperatively and postoperatively.
Change in Pediatric Voice-Related Quality of Life Scores | Preoperative, 1 month postoperative, and 3 months postoperative
  Voice-related quality of life will be evaluated using the Pediatric Voice-Related Quality of Life (PVRQOL) questionnaire. Scores range from 0 to 100, with higher scores indicating better voice-related quality of life. The validated Turkish version will be used.

CONTACTS AND LOCATIONS:
Overall Officials: DERYA CEBECİ, MD, Principal Investigator — Gaziosmanpaşa Training and Research Hospital, Department of Otolaryngology
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared outside of the research team due to the sensitive nature of pediatric patient data and privacy considerations.

REFERENCES:
- [Background] An evaluation of the effects of adenoidectomy on voice and speech function in children. Medine Kara, Kayhan Öztürk, Bedri Özer. Kulak Burun Bogaz Ihtis Derg 2013;23(4):225-231. doi: 10.5606/kbbihtisas.2013.09476.
- [Background] Adenotonsillektominin Akustik, Algısal ve Aerodinamik Ses Parametrelerine Etkisi. Beyhan Yılmaz, Engin Sengul, Musa Özbay, Salih Bakır. Dicle Tıp Dergisi /Dicle Medical Journal 2016; 43 (2): 333-338. doi: 10.5798/diclemedj.0921.2016.02.0691
- [Background] Inja RR, Paul RR, Varghese L, Santosh S, Sebastian T, Mathews SS. Voice Change Following Adenotonsillectomy in Pediatric Population: Myth or Reality?-A Pilot Study. Indian J Otolaryngol Head Neck Surg. 2019 Oct;71(Suppl 1):574-579. doi: 10.1007/s12070-018-1412-6. Epub 2018 Jun 4. PMID 31742023